CLINICAL TRIAL: NCT05606718
Title: Dapagliflozin Effect on FunctiOnal Mitral Regurgitation and Myocardial Remodeling
Acronym: DEFORM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, Prof, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEFORM trial
Record Dates: First submitted 2022-10-30; First posted 2022-11-07 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Functional Mitral Regurgitation
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dapagliflozin group (Experimental): GDMT and dapagliflozin 10mg once daily
  Interventions: Drug: Dapagliflozin; Other: guideline-directed medical therapy (GDMT)
- control group (Active Comparator): GDMT only
  Interventions: Other: guideline-directed medical therapy (GDMT)

INTERVENTIONS:
Drug: Dapagliflozin — dapagliflozin 10mg once daily for 3 months after randomization
  Arms: dapagliflozin group
Other: guideline-directed medical therapy (GDMT) — guideline-directed medical therapy (GDMT)

SUMMARY:
Functional mitral regurgitation (FMR) leads to various adverse outcomes. Cardiac remodeling (CR) and myocardial fibrosis (MF) are closely related to FMR, forming a vicious circle of CR-FMR-MF and resulting in the end-stage heart failure (HF). The optimal therapeutic strategies of FMR require to effectively break the vicious circle of CR-FMR-MF and still remain full of controversy, especially in the appropriate selection of patients suitable for transcatheter treatment. Regardless, adequate guideline-directed medical therapy (GDMT) is always the most important therapy of FMR. Currently GDMT for FMR included β-blockers, renin-angiotensin system (RAS) inhibitors and mineralocorticoid receptor antagonists (MRA). Dapagliflozin, a sodium-glucose cotransporter-2 inhibitor, have been proven to be effectively in reducing cardiovascular death and worsening HF in HF patients. However, there is still no evidence support the use of SGLT2i in FMR therapy due to the lack of relevant clinical trial. The DEFORM trial aims to assess the efficacy of dapagliflozin in reducing the extent of mitral regurgitation and myocardial fibrosis in FMR patients. DEFORM trial is a multi-center, prospective, randomized, parallel controlled, investigator-initiated trial enrolling a planned 98 FMR patients. Patients will be randomly assigned in a 1:1 ratio to either dapagliflozin 10mg once daily for 3 months or placebo. The primary outcome is the change in effective regurgitant orifice area (EROA) of mitral regurgitation measured by echocardiography. Secondary end-points include change change in regurgitant volume (RV), left ventricular end-systolic volume (LVESV), left ventricular end-diastolic volume (LVEDV) (echocardiography), change in NT-proBNP levels and occurrence of major adverse cardiac events (MACEs).

DETAILED DESCRIPTION:
Inclusion criteria:

* Patients aged >18 years and <90 years
* LVEF<60% and EROA of mitral regurgitation≥0.2cm2 on echocardiography
* The structure of mitral valve leaf and chordae tendineae is normal
* Patients have received GDMT for FMR including a stable, optimized dose of β-blocker and RAAS inhibitors for at least 2 weeks
* No intravenous anti-heart failure drugs used for the past 2 weeks
* Written informed consent

Exclusion criteria:

* Allergic to dapagliflozin, or angioedema
* Already taking dapagliflozin or other SGLT2 inhibitors
* Presence of primary structural damage to the mitral valve, such as rheumatic heart disease, mitral valve prolapses
* Non-dialysis chronic kidney disease (CKD) patients with eGFR <30ml/min/1.73m2 or dialysis patients
* Acute myocardial infarction and acute myocarditis occurred within 3 months
* Revascularization procedure, CRT, TMVR, surgical valve repair or replacement were performed or planed 3 months before or after enrollment
* Combining significant aortic valve diseases (moderate or severe regurgitation or stenosis)
* Combining hyperthyroidism while thyroid function has not returned to normal
* Pregnant or lactation women

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years and <90 years
* LVEF<60% and EROA of mitral regurgitation≥0.2cm2 on echocardiography
* The structure of mitral valve leaf and chordae tendineae is normal
* Patients have received GDMT for FMR including a stable, optimized dose of β-blocker and RAAS inhibitors for at least 2 weeks

Exclusion Criteria:

* Allergic to dapagliflozin, or angioedema
* Already taking dapagliflozin or other SGLT2 inhibitors
* Presence of primary structural damage to the mitral valve, such as rheumatic heart disease, mitral valve prolapses
* Non-dialysis chronic kidney disease (CKD) patients with eGFR <30ml/min/1.73m2 or dialysis patients
* Acute myocardial infarction and acute myocarditis occurred within 3 months
* Revascularization procedure, CRT, TMVR, surgical valve repair or replacement were performed or planed 3 months before or after enrollment
* Combining significant aortic valve diseases (moderate or severe regurgitation or stenosis)
* Combining hyperthyroidism while thyroid function has not returned to normal
* Pregnant or lactation women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
EROA of FMR | 3 months
  Change in EROA of mitral regurgitation evaluated by echocardiography from baseline to 12 weeks follow-up

SECONDARY OUTCOMES:
cardiac structure | 3 months
  Change in RV measured by echocardiography from baseline to 12 weeks follow-up
MACE | 3 months
  Occurrence of MACE in 12 weeks follow-up
cardiac function | 3 months
  Change in serum NT-proBNP levels from baseline to 12 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Zhuang, Dr, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (3):
- China (3):
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University Yuedong Hospital, Meizhou, Guangdong

IPD SHARING:
Plan to Share IPD: No